CLINICAL TRIAL: NCT01661309
Title: To Critically Investigate and Evaluate Supplementary Vitamin B12 Effects on Elevated Homocysteine Levels of Vegetarians, Who May Have a Resultant Susceptibility to Hyperhomocysteinemia Related Diseases.
Brief Title: Supplementary Vitamin B12 Effects on Elevated Homocysteine Levels of Vegetarians - Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of West London (Other)
Responsible Party: Principal Investigator, Derek Obersby, PhD Student, University of West London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Methylcobalamin
Record Dates: First submitted 2012-08-06; First posted 2012-08-09 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Vitamin B12 Deficiency
Keywords: Hyperhomocysteinemia; Methylcobalamin; Cardiovascular disease; Plasma total homocysteine; Vegetarians
MeSH Terms: conditions — Vitamin B 12 Deficiency; Hyperhomocysteinemia; Cardiovascular Diseases | interventions — mecobalamin; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inactive lozenge (Placebo Comparator): Inactive lozenge containing 2mg sucrose dissolved in the mouth taken after a meal every other day for 16 weeks
  Interventions: Dietary Supplement: Inactive lozenge; Dietary Supplement: Methylcobalamin
- Methylcobalamin (Experimental): Methylcobalamin 1mg lozenge dissolved in the mouth following a meal taken every other day for 16 weeks.
  Interventions: Dietary Supplement: Inactive lozenge; Dietary Supplement: Methylcobalamin

INTERVENTIONS:
Dietary Supplement: Inactive lozenge — Manufactured to mimic 1mg methylcobalamin lozenge
Dietary Supplement: Methylcobalamin — Aimed at reducing plasma tHcy.
  Other Names: Vitamin B12

SUMMARY:
Vegetarians are known to be deficient in vitamin B12, due to a lack or absence of dietary animal produce, which can elevate homocysteine. There is strong evidence indicating that elevated plasma total homocysteine (tHcy) is a contributor to chronic conditions, such as primary cardiovascular disease (CVD). The study hypothesis is: There will be a significant decrease in plasma tHcy of vegetarians following the intervention by supplementary vitamin B12 (of the methylcobalamin type) and this will lead to a reduction of the risk of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Having a plasma tHcy >10 micromol/L
* Not suffering from conditions as described in exclusion criteria.
* Vegetarian for at least one year.
* Not participating in a weight reducing diet.
* Not consuming regularly vitamin B12 supplements.
* Give written consent to participate in clinical trial and be fluent in English language.

Exclusion Criteria:

* Having a plasma tHcy less or equal to 10 micromol/L.
* Suffering from pernicious anemia or other vitamin B12 deficiency disease.
* Undergone bowel surgery or suffer from gastrointestinal disease.
* Pregnant, lactating or trying to conceive.
* Smoker.
* Alcohol intake regularly greater than official recommended daily units (i.e. 2 units female, 3 units male).
* Consume large amounts of caffeine (regular consumption of >4 cups of strong tea or coffee per day).
* Use of medications known to influence nutritional status.
* Have genetic metabolic disease.
* Suffer from renal failure, diabetes, thyroid disease, cardiovascular disease, dementia or cancer.
* Have a known blood-borne infection (e.g. Hepatitis or HIV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Reduction of plasma total homocysteine of vegetarians | 16 weeks per participant

SECONDARY OUTCOMES:
Improvement in systolic and diastolic blood pressure | 16 weeks per participant

OTHER OUTCOMES:
Improvement in body mass index | 16 weeks per participant

CONTACTS AND LOCATIONS:
Overall Officials: Amalia A Tsiami, PhD, Study Director — University of West London; David C Chappell, PhD, Study Director — University of West London
Locations (1):
- University of West London, London, Middlesex, United Kingdom